CLINICAL TRIAL: NCT02721797
Title: Origins and Impact of EDS in Connective Tissues and Skin
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 15/0438
Record Dates: First submitted 2016-03-02; First posted 2016-03-29 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Ehlers-Danlos Syndrome
Keywords: hypermobility; collagen; joint; hyperflexation
MeSH Terms: conditions — Ehlers-Danlos Syndrome | interventions — Orthopedic Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collagen in skin, tendon, ligament, vaginal tissue, uterine tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Skin: Patients with EDS diagnosis having surgery, have debrided skin retained for this research
  Interventions: Procedure: Orthopaedic & Gynaecology surgery
- Tendon: Patients with EDS diagnosis having surgery, have debrided tendon retained for this research
  Interventions: Procedure: Orthopaedic & Gynaecology surgery
- Uterine tissue: Patients with EDS diagnosis having surgery, have debrided uterine tissue retained for this research
  Interventions: Procedure: Orthopaedic & Gynaecology surgery
- Vaginal tissue: Patients with EDS diagnosis having surgery, have debrided vaginal tissues retained for this research
  Interventions: Procedure: Orthopaedic & Gynaecology surgery
- Ligaments: Patients with EDS diagnosis having surgery, have debrided ligaments retained for this research
  Interventions: Procedure: Orthopaedic & Gynaecology surgery

INTERVENTIONS:
Procedure: Orthopaedic & Gynaecology surgery — Patients will have the surgery they require for their treatment. During surgery, debrided tissues will be retained for research. No treatment plans will be altered for this research.

SUMMARY:
Ehlers-Danlos Syndrome (EDS) is an inherited disease of collagen, found in connective tissues, such as skin. EDS patients suffer from joint and skin problems (skin hyperextensibility, joint hypermobility) along with a large range of other disorders, including, delayed wound healing with atrophic scarring, easy bruising, tissue fragility, gastrointestinal and gum problems. There are many different types of EDS, with different mechanisms of action, and not all of these are well understood. This study will used advanced microscopy techniques called atomic force microscopy (AFM) and scanning electron microscopy (SEM) to analyse the changes in collagen as a result of EDS, compared to normal collagen. These changes will be viewed at the micron and nanoscale level (between 1,000 to 100,000 x magnification), and will focus on the differences in collagen construction through a process called cross-linking. These changes could potentially help clinicians understand the root cause of EDS symptoms, and provide a deeper knowledge of cross-linking disorders in collagen. Increasing our knowledge of how collagen is affected in EDS patients, may lead to improved treatment options for patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+) patients requiring elective surgery as part of their treatment plan who fulfil the Brighton criteria for Joint Hypermobility Syndrome (JHS)/EDS hypermobility type with significant joint hypermobility (Beighton score of 6 and above) and /or have evidence of significant connective tissue weakness, or rectal/vaginal prolapse

Exclusion Criteria:

* Patients with insufficient ability in English to give informed consent, if a translator is not present.
* Patients with severe developmental disorders, precluding their consent for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be identified from screening of all new and existing Hypermobility, Orthopaedics and Gynaecology clinics at UCLH and invited to participate in the study. The appropriate information sheet will be given to the patients who have been identified for elective surgery as part of their treatment plan and meeting the inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Histological changes in EDS compared with healthy collagen using light microscopy after staining | 1-5 years
  Light microscopy will be qualitatively used to observe colour changes after staining between healthy and EDS collagen
Collagen morphological changes in EDS compared with healthy collagen using AFM and SEM | 1-5 years
  AFM and SEM will be used to qualitatively observe changes in orientation in collagen.
Collagen topographical changes in EDS compared with healthy collagen using AFM and SEM | 1-5 years
  AFM and SEM will be used to observe changes in length, width and height of healthy and EDS collagen, as well as D-band length. This will be measured in meters (nm).

SECONDARY OUTCOMES:
Collagen Young's modulus changes in EDS compared with healthy collagen using AFM | 1-5 years
  AFM will be used to calculate the Young's (elastic) modulus of the EDS and healthy collagen. This will be measured in Pascals (GPa).
Collagen nanoscale adhesion changes in EDS compared with healthy collagen using AFM | 1-5 years
  AFM will be used to calculate the changes in adhesion force of the EDS and healthy collagen. This will be measured in Newtons (nN).
  Quantitative outcomes: changes in Young's (elastic) modulus, changes in adhesion force, changes in single molecule pulling force
Collagen nanoscale single molecule pulling force in EDS compared with healthy collagen using AFM | 1-5 years
  AFM will be used to calculate the changes in pulling force of single molecules of EDS and healthy collagen. This will be measured in Newtons (nN).

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Kazkaz, Principal Investigator — UCLH; Laurent Bozec, Principal Investigator — UCL; Adam Strange, Principal Investigator — UCL; Rodney Graham, Principal Investigator — UCL; Susan Parekh, Principal Investigator — UCLH
Locations (1):
- University Collage Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No data will be shared outside of this research